CLINICAL TRIAL: NCT01238042
Title: A Pilot Study To Determine The Maximum Range of Light Doses At Two HPPH Doses With Acceptable Normal Tissue Toxicity For PDT Treatment Of High Grade Dysplasia,CIS or Early Adenocarcinoma In Barrett's Esophagus
Brief Title: Study To Determine The Maximum Range of Light Doses At Two HPPH Doses With Acceptable Normal Tissue Toxicity For PDT Treatment Of High Grade Dysplasia,CIS or Early Adenocarcinoma In Barrett's Esophagus
Status: Completed | Phase: Phase 1 | Type: Interventional
Sponsor: Roswell Park Cancer Institute (Other)
Responsible Party: Sponsor
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: RP 02-18
Record Dates: First submitted 2010-11-01; First posted 2010-11-10 (Estimated); Last update posted 2014-12-02 (Estimated); Status verified 2014-12

CONDITIONS: Barrett's Esophagus; CIS; HGD
MeSH Terms: conditions — Barrett Esophagus | interventions — 2-(1-hexyloxyethyl)-2-devinyl pyropheophorbide-a

STUDY DESIGN:
Oversight: Data Monitoring Committee: Yes

ARMS (1):
- Light Dose Escalation (Experimental): Light Dose escalated from 150 joules/cm to 200 joules/cm
  Interventions: Drug: HPPH

INTERVENTIONS:
Drug: HPPH — 3mg/m2 or 4 mg/m2 at light doses of 150, 175 and 200 joules/cm

SUMMARY:
Patient's with High Grade Dysplasia, Carcinoma in situ or Early Adenocarcinoma in Barrett's Esophagus are injected with HPPH and one day later are endoscopically treated with light from a laser.

ELIGIBILITY:
Inclusion Criteria:

* Patient must have biopsy proven high-grade (severe)dysplasia, carcinoma-in-situ or early stage adenocarcinoma
* Patient may have received prior therapy; e.g.Nd-YAG laser, radiation therapy or chemotherapy. At least one-month must have elapsed between prior treatments and PDT
* Tumors (HGD/CIS or early adenocarcinoma) can be primary or recurrent, Stage 0 or I N0M (any)
* Patients must have no contraindication to endoscopy
* Male or female patients must be 18 years old or older. Female patients must not be pregnant and must be practicing a medically acceptable form of birth control or be sterile or post-menopausal. A Pregnancy test is required and must be negative.
* Patients must sign an Informed Consent according to FDA guidelines and be acceptable to the RPCI IRB
* Patients must have a Karnofsky status 50 or above.
* Patients with early invasive adenocarcinoma will be included only if they are considered poor surgical risks, have failed or refused XRT/chemo, or refused surgery.
* If the patients has had cancer other than non-melanoma skin cancer, their treating physician must deem them disease-free.

Exclusion Criteria:

* Patients with tumors of grade greater than T-1.
* Porphyria or hypersensitivity to porphyrin or porphyrin-like compounds
* WBC<4000; platelet count<100,000; prothrombin times 1.5 times above upper normal limit.
* Patients with impaired renal and/or hepatic function (total serum bilirubin > 3.0 mg/d, serum creatinine>3 mg%, alkaline phosphatase (hepatic) or SGOT> 3 times the upper normal limit.
* Patients on concurrent chemotherapy or radiation therapy will be excluded as well as those having received prior treatment for the esophageal cancer within 4 weeks of enrollment.

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 18 (Actual)
Dates: Start 2003-03; Primary Completion 2004-10 (Actual); Study Completion 2014-11 (Actual)

PRIMARY OUTCOMES:
Optimal Light Dose | 24 hours
  Using toxicity to normal surrounding tissue as a determinant and using two HPPH doses of PDT in HGD, CIS or early adenocarcinoma in Barrett's esophagus, to determine the optimal light dose at each HPPH dose

SECONDARY OUTCOMES:
Toxicity to normal surrounding tissue | 24 hours
  To determine the tocixity to normal surrounding tissue of treating at approximately 24 hours(21-26hr) post injection of HPPH
Comparing HPPH to Photofrin | 5 years
  To determine the length of time of cutaneous photosensitivity of HPPH compared to historical data on Photofrin
Effect of injection | 24 hours
  To determine the effect of a 24 hours interval between injection of HPPH and light treatment
Efficacy of Treatment | 5 years
  A secondary objective is to determine efficacy of treatment at each set of paraments, i.e. ability to completely resolve the CIS, HGD or early cancer.
Resolve Barrett's mucosa | 5 years
  An Additional secondary objective is to determine ability of PDT to resolve the Barrett's mucosa

CONTACTS AND LOCATIONS:
Overall Officials: Hector Nava, MD, Principal Investigator — Roswell Park Cancer Institute
Locations (1):
- Roswell Park Cancer Institute, Buffalo, New York, United States